CLINICAL TRIAL: NCT00618553
Title: The Efficacy of Pulmonary Rehabilitation in Improving Surgical Eligibility for Lung Resection
Brief Title: Effect of Pulmonary Rehabilitation on Surgical Outcomes in the Cancer Setting
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-0063; NCI-2012-01749 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-01-28; First posted 2008-02-20 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Pulmonary Rehabilitation; Questionnaire; Survey; Lung Function; Quality of Life
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): Pulmonary Rehabilitation - Rehabilitation treatment given over about 3-4 weeks. Questionnaire regarding quality-of-life that lasts about 30 minutes.
  Interventions: Other: Questionnaire; Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Questionnaire — Questionnaire regarding quality-of-life that lasts about 30 minutes.
  Other Names: Survey
Behavioral: Pulmonary Rehabilitation — Rehabilitation treatment given over about 3-4 weeks.

SUMMARY:
The goal of this clinical research study is to see if pulmonary rehabilitation can improve patients' lung function, which would increase their chances of becoming eligible for surgery. The health of pulmonary rehabilitation participants after surgery will also be examined.

DETAILED DESCRIPTION:
Pulmonary rehabilitation is a process that is designed to improve patients' lung function, muscular conditioning, exercise performance, and overall quality of life.

Study activities include exercise training, patient and family education, and psychosocial and behavioral counseling provided by a healthcare team.

Rehabilitation plans will vary patient by patient based on the results of the following tests:

* Blood (1-3 tablespoons) will be drawn for routine tests.
* You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart).
* You will have an X-ray of your chest.
* You will have a Pulmonary Function Test. For this test, you will be asked to breathe in several different ways while you have a mouthpiece in your mouth to test your lung function.

Study Visits:

If you choose to take part in this study, you will have 3-4 weeks of pulmonary rehabilitation. During the 3-4 week period, you will have 9-12 study visits that will last about 90 minutes each. The following tests and procedures will be performed:

6-Minute Walk Test:

To perform the 6-minute walk test, you will walk as far as possible around cones on a flat indoor course that is about 40 yards long. You will walk at your own pace and can take breaks at any time. After 6 minutes, the study staff will check the total distance you have walked. Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be measured before and after the walk. Your oxygen saturation levels will be monitored throughout the test. You will wear a small clip on your finger that will send the oxygen saturation data to a small computer.

Oxygen Consumption Test:

An oxygen consumption study will help the doctor determine how well your heart and lungs work while you exercise. You will be asked to pedal on a bicycle that does not move, while wearing a mouthpiece to measure the amount of oxygen you take in. Wires will be placed on your chest to monitor your heart activity, and a blood pressure cuff will be placed on your arm to monitor your blood pressure.

The amount of exercise you can do will be measured by increasing the resistance you pedal against. You should continue pedaling until you become short of breath or too tired to keep going. You may stop exercising at any time if you become very uncomfortable or experience dizziness, chest pains, and/or shortness of breath.

During or after the oxygen consumption test, blood (about 2 teaspoons) may be drawn to measure the amount of oxygen in your blood.

If you live outside of the Houston area, you will be referred to a pulmonary rehabilitation program in your local area. Any records from the outside pulmonary rehabilitation facility will be given to the study staff after the study is completed. You will have your follow-up visits (described below) at M. D. Anderson.

Follow-up Visits:

Your health status will be checked at 1 and 3 months after your last study visit if you do not have surgery, or 1 and 3 months after your surgery. At these follow-up visits, the following tests and procedures will be performed:

* You will have a 6-minute walk test, a Pulmonary Function Test, and an Oxygen Consumption Test.
* You will be asked to fill out a quality-of-life questionnaire that should take about 30 minutes to complete.
* You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation).
* An echocardiogram will be done on a patient-by patient basis. An echocardiogram uses sound waves to make pictures of your heart, which helps show how well your heart pumps blood. You will be asked to lie on your left side while a technician places a probe with gel on your chest to create images of your heart to determine the function and size.

Long-term Follow-up:

The research staff may contact you by phone regarding your health status. Patients who have lung surgery may be contacted by phone or have their medical records reviewed during the course of 30 days after surgery or during hospitalization for surgery (hospitalization may last more than 30 days).

This is an investigational study. Using pulmonary rehabilitation to try to improve patients' lung function is considered experimental. At this time, it is being done in research only. Up to 75 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with anatomically resectable lung tumors who are deemed surgically inoperable based on preoperative pulmonary function testing FEV1 < 80% pred; DLCO < 80% pred; FEV1ppo < 40% pred; DLCO ppo < 40% pred AND VO2 peak < 60% predicted or < 15 ml/kg/min.
2. Patients deemed surgically inoperable based on poor performance status (ECOG score 2-3)
3. Any non-pulmonary co-morbidity must be stable according to institutional guidelines.

Exclusion Criteria:

1. Previously reported severe pulmonary hypertension (pulmonary artery systolic pressure > 60 as determined by echocardiogram), refractory cor pulmonale (as manifested by right ventricular dilatation or dysfunction by echocardiogram)
2. Previously reported exercise-induced syncope, angina, palpitation, arrhythmia, hypotension (drop of 20% of systolic/diastolic from baseline)
3. History of severe congestive heart failure (NYHA class 3 and 4) refractory to medical management, (LVEF < 40% by echocardiogram).
4. Bone metastasis
5. Active psychiatric illness that could interfere with treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-01-28 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Success (conversion from ineligible to eligible status for lung resection following Pulmonary rehabilitation (PR)) | Baseline and post treatment (following 3-4 weeks of PR)

SECONDARY OUTCOMES:
Examine health of pulmonary rehabilitation participants after surgery. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Vickie Shannon, BS,MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org